CLINICAL TRIAL: NCT00004102
Title: A Phase II Trial of Eloxatin in Combination With 5-Fluorouracil and Leucovorin in Patients With Advanced Colorectal Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067321; P30CA016087 (NIH); NYU-9863; SANOFI-EFC7132; NCI-G99-1593
Record Dates: First submitted 1999-12-10; First posted 2004-04-12 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Leucovorin may increase the effectiveness of fluorouracil by making tumor cells more sensitive to the drug.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of oxaliplatin, fluorouracil, and leucovorin in treating patients who have colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the quantitative and qualitative toxicities of oxaliplatin combined with fluorouracil and leucovorin calcium in patients with advanced adenocarcinoma of the colon or rectum.

OUTLINE: Patients receive leucovorin calcium IV over 10-20 minutes followed within 10 minutes by fluorouracil IV bolus on days 1, 8, 15, 29, 36, and 43. Patients receive oxaliplatin IV over 2 hours prior to leucovorin calcium and fluorouracil on days 1, 15, 29, and 43. Treatment repeats every 8 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may receive additional courses upon approval by the sponsor. Patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced adenocarcinoma of the colon or rectum No prior systemic chemotherapy OR Adjuvant chemotherapy only, completed 6 months prior to study and with subsequent development of recurrent disease At least 1 bidimensionally measurable lesion No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL (no greater than 5.0 mg/dL if due to intrahepatic biliary obstruction not amenable to biliary decompression, if approved by the protocol investigator) SGOT no greater than 4 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No myocardial infarction within the past 6 months No congestive heart failure Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No neurologic disease No active or uncontrolled infection No other malignancy within the past 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix No medical or psychiatric disorders that would prevent compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for malignant disease Surgery: Recovered from any prior surgery Other: At least 30 days since other prior investigational agent No other concurrent investigational agents No concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01; Primary Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Hochster H, Chachoua A, Speyer J, Escalon J, Zeleniuch-Jacquotte A, Muggia F. Oxaliplatin with weekly bolus fluorouracil and low-dose leucovorin as first-line therapy for patients with colorectal cancer. J Clin Oncol. 2003 Jul 15;21(14):2703-7. doi: 10.1200/JCO.2003.02.071. PMID 12860947